CLINICAL TRIAL: NCT01714362
Title: Prediction of Oculocardiac Reflex in Relationship to Autonomic Nervous System Activity, Mesured With the Use of ECG HRV Analysis.
Brief Title: Autonomic Nervous System Activity and Oculocardiac Reflex.
Status: Completed | Type: Observational
Sponsor: Medical University of Gdansk (Other)
Responsible Party: Principal Investigator, Magdalena Wujtewicz, assistant professor, Medical University of Gdansk
Other Study IDs: GUMed-Ow-003
Record Dates: First submitted 2012-10-23; First posted 2012-10-25 (Estimated); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Bradycardia During Pulling of Eyeball
Keywords: oculocardiac effect; bradycardia; HRV
MeSH Terms: conditions — Bradycardia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Pulling the eyeball during ophthalmic surgery provokes decrease in heart rate. This phenomenon is called oculocardiac reflex. In some patients asystole may occur. Other cardiac features of this reflex include hypotension, dysrhythmias, atrioventricular block. These cardiovascular disturbances may lead to decreased perfusion and ischemia of vital organs. Patients with existing cardiovascular disease are in risk of complications. Cardiovascular system is mainly innervated with autonomic nervous system (ANS). Sympathetic/parasympathetic activity may be determined by Heart Rate Variability (HRV). HRV analysis based on short 5 minutes electrocardiography has been found useful for prediction of hypotension and bradycardia during induction of general anaesthesia and during spinal block. The aim of this study is to verify whether it is possible to predict oculocardiac reflex with the use of HRV analysis for ANS activity assessment, measured prior to the ophthalmic surgery.

ELIGIBILITY:
Inclusion Criteria:

* planned surgery
* over 18 years of age
* surgery under general anaesthesia

Exclusion Criteria:

* urgent surgery
* under 18 years of age and over 65
* patients with generalised, nontreated disease
* patients receiving beta blockers or calcium channel blocker
* diabetic patients
* patients operated under peri or retrobulbar anaesthesia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients operated bacause of retinal pathology
Sampling Method: Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2009-10 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
oculocardiac reflex occurence in relation to autonomic system activity | perioperatively - about 2 hours

CONTACTS AND LOCATIONS:
Overall Officials: Magdalena A Wujtewicz, MD PhD, Principal Investigator — Department of Ophthalmology, Mediacal University of Gdansk, Gdansk, Poland
Locations (1):
- Medical University of Gdansk, Gdansk, Poland

REFERENCES:
- [Derived] Wujtewicz M, Twardowski P, Jasinski T, Raczynska D, Owczuk R. Prediction of the Occurrence of the Oculocardiac Reflex Based on the Assessment of Heart Rate Variability. An Observational Study. Ophthalmol Ther. 2022 Oct;11(5):1857-1867. doi: 10.1007/s40123-022-00549-0. Epub 2022 Aug 1. PMID 35913657